CLINICAL TRIAL: NCT00980512
Title: Community Implementation of KEEP: Fidelity and Generalization of Parenting
Acronym: KEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Dr. Joseph M. Price, PI, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH060195 (NIH); R01MH060195 (NIH); 2R01MH060195-06A1 (NIH); DSIR 84-CTP
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Behavior Problems
Keywords: behavior problems; parent training; foster care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Training (Experimental): Parent Training of foster parents
  Interventions: Behavioral: Parent Training
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Parent Training — 16 weeks of parent training led by trained group facilitator
  Other Names: Parent Management Training
  Arms: Parent Training

SUMMARY:
The primary goal of this study is to examine the fidelity and generalization of parenting effects of the KEEP foster parent training intervention as it is being delivered within a child welfare system of care by a community mental health provider.

DETAILED DESCRIPTION:
The primary goal of this study is to utilize this opportunity as a real-world platform for addressing three key questions that need to be answered prior to wide-scale implementation of the KEEP intervention. First, do the effects of the KEEP parent training generalize (concurrently) to other children currently in foster and kin intervention homes and lead to reductions in overall levels of behavior problems? Second, does the KEEP intervention continue to have effects after the completion of the intervention and generalize (temporally) to new children who enter the homes of these families at a later point in time? Finally, as the KEEP intervention is being implemented by a community agency in a real-world system of care, can the intervention be delivered and maintained in a manner that preserves the goals and quality of the intervention?

Children in foster care, between the ages of 5 and 12, will be randomly assigned to one of two conditions - the KEEP intervention or a "services as usual" condition. In the KEEP intervention condition, foster and kin caregivers will participate in 16 weekly group meetings. Outcomes to be assessed include child problem behavior (of the focal child and other children in the household), child functioning, parental stress, family functioning, use of mental health services, child placement changes (e.g., reunification with biological parents, move to another foster home), and foster parent retention rates. In addition, for a year following the completion of the intervention, new children entering the home of foster/kin caregiver will be included in the assessments, along with the impact of these additional children on parental stress and family functioning. Finally, several dimensions of intervention fidelity (e.g., facilitator adherence and group engagement) will be assessed and examined in relation to child, family, and system outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any child between ages 5 and 12 in relative or non-relative foster care

Exclusion Criteria:

* Only medically fragile children

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction in child behavior problems as assessed by the Parent Daily Report (PDR) | Baseline, 6-months, 12-months, 18-months

SECONDARY OUTCOMES:
Placement Disruptions from Foster Placement | 6-month, 12-month, 18-month

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Price, Ph.D., Principal Investigator — San Diego State University & Child and Adolescent Services Research Center
Locations (1):
- Child and Adolescent Services Research Center, San Diego, California, United States

REFERENCES:
- [Background] Chamberlain P, Price J, Leve LD, Laurent H, Landsverk JA, Reid JB. Prevention of behavior problems for children in foster care: outcomes and mediation effects. Prev Sci. 2008 Mar;9(1):17-27. doi: 10.1007/s11121-007-0080-7. Epub 2008 Jan 10. PMID 18185995
- [Background] Price JM, Chamberlain P, Landsverk J, Reid JB, Leve LD, Laurent H. Effects of a foster parent training intervention on placement changes of children in foster care. Child Maltreat. 2008 Feb;13(1):64-75. doi: 10.1177/1077559507310612. PMID 18174349
- [Background] Chamberlain P, Price J, Reid J, Landsverk J. Cascading implementation of a foster and kinship parent intervention. Child Welfare. 2008;87(5):27-48. PMID 19402358
- See also: Child and Adolescent Services Research Center — http://casrc.org